CLINICAL TRIAL: NCT00884312
Title: An Open-Label, Single-Arm, Phase 2 Study of Extended Carfilzomib Therapy in Subjects Previously Enrolled in Carfilzomib Treatment Protocols
Brief Title: A Study of Extended Carfilzomib Therapy for Patients Previously Enrolled in Carfilzomib Treatment Protocols
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-010; 20130394 (Other: Amgen Study ID)
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Multiple Myeloma; Solid Tumors
Keywords: Multiple myeloma; proteasome; Hematological; carfilzomib; PR-171
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib (Experimental): Participants received carfilzomib administered intravenously, using the same method, frequency, and dose level as in the last cycle of the participant's previous carfilzomib study. Treatment was continued until confirmation of disease progression, diagnosis of new malignancy, unacceptable toxicity, investigator discretion, voluntary withdrawal, or commercial availability of carfilzomib.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib dose levels ranged from 11 to 27 mg/m² for 2- to 10-minute infusions and 36 to 56 mg/m² for 30-minute infusions. Carfilzomib doses were administered on days 1, 2, 8, 9, 15, and 16 of a 28-day cycle. Dose level reduction to a minimum dose of 11 mg/m² for toxicity was permitted.
  Other Names: PR-171; PR171; Kyprolis®

SUMMARY:
This is a multi-center, open-label, Phase 2 study of carfilzomib to monitor the safety and efficacy of long-term or continuing carfilzomib therapy for patients who previously completed a primary carfilzomib treatment study.

ELIGIBILITY:
Inclusion Criteria:

1. Previous completion of a carfilzomib study within 90 days prior to first dose of maintenance study drug.
2. Disease Assessments performed within 30 days prior to first dose of maintenance study drug.
3. Written informed consent in accordance with federal, local, and institutional guidelines
4. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test, with a sensitivity of at least 50 mIU/mL, within 3 days prior to first dose of maintenance study drug.
5. Subjects must agree to adhere to the study visit schedule and other study requirements and receive outpatient treatment and laboratory monitoring at the institution that administers the drug.

Exclusion Criteria:

1. Administration of an intervening chemotherapy between the time of previous carfilzomib study termination and first dose of maintenance study drug.
2. Pregnant or lactating females
3. Diagnosis of a new malignancy of a different tumor type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-04-09 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- United States (21):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope National Medial Center, Duarte, California
  - University of California Medical Center, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology Cancer Center, Austin, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Northwest Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (2):
  - University of Toronto, Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 23 centers in the United States and Canada from April 2009 to May 2017.
Groups:
- Solid Tumors: Participants with solid tumors received carfilzomib administered intravenously, using the same method, frequency, and dose level as in the last cycle of the participant's previous carfilzomib study. Treatment was continued until confirmation of disease progression, diagnosis of new malignancy, unacceptable toxicity, investigator discretion, voluntary withdrawal, or commercial availability of carfilzomib.
- Multiple Myeloma: Participants with multiple myeloma received carfilzomib administered intravenously, using the same method, frequency, and dose level as in the last cycle of the participant's previous carfilzomib study. Treatment was continued until confirmation of disease progression, diagnosis of new malignancy, unacceptable toxicity, investigator discretion, voluntary withdrawal, or commercial availability of carfilzomib.
Period: Overall Study
Arm/Group | Solid Tumors | Multiple Myeloma
Started | 9 | 92
Received Treatment | 9 | 91
Completed (Completed final visit) | 7 | 67
Not Completed | 2 | 25
Not completed — Non-fatal Progressive Disease | 0 | 8
Not completed — Fatal Progressive Disease | 0 | 1
Not completed — Non-fatal Adverse Event | 1 | 0
Not completed — Fatal Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Other | 0 | 4
Not completed — Did Not Receive Study Drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of carfilzomib after enrollment in PX-171-010.
Groups:
- Total: Total of all reporting groups
Arm/Group | Solid Tumors | Multiple Myeloma | Total
Number analyzed (Participants) | 9 | 91 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.75) | 63.2 (9.82) | 63.0 (10.05)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 5 | 47 | 52
  ≥ 65 years | 4 | 44 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 38 | 44
  Male | 3 | 53 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 71 | 80
  Black | 0 | 11 | 11
  Hispanic | 0 | 5 | 5
  Asian/Pacific Islander | 0 | 4 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 6 | 39 | 45
    1 (Restricted but ambulatory) | 3 | 42 | 45
    2 (Ambulatory but unable to work) | 0 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Peripheral Neuropathy
Description: Participants with peripheral neuropathy or peripheral neuropathy-related adverse events, including hypoaesthesia, paraesthesia, dysaesthesia, and neuropathic pain.
Time Frame: From first dose of study drug to 30 days after the last dose; median duration of treatment was 14 weeks for participants with solid tumors and 44 weeks for participants with multiple myeloma.
Population: All participants who received at least 1 dose of carfilzomib after enrollment in PX-171-010.
Measure: Number; unit: participants
Arm/Group | Solid Tumors | Multiple Myeloma
Number analyzed (Participants) | 9 | 91
participants | 1 | 15

2. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were assigned a severity grade using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grading scale version 3.0.
  Per protocol, adverse events were collected if they led to dose modification or dose discontinuation, were grade ≥ 3 or serious, or were events of peripheral neuropathy (any grade).
  A serious AE is one that met one or more of the following criteria:
  * Death
  * Life threatening
  * Required inpatient hospitalization or prolongation of an existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * A congenital anomaly/birth defect in the offspring of an exposed subject
  * Important medical events that, based upon appropriate medical judgment, jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes above.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of carfilzomib after enrollment in PX-171-010.
Measure: Number; unit: participants
Arm/Group | Solid Tumors | Multiple Myeloma
Number analyzed (Participants) | 9 | 91
participants
  Any adverse event | 7 | 84
  Adverse event ≥ grade 3 | 5 | 66
  Serious adverse events | 5 | 57
  Fatal adverse events | 1 | 7
  AE leading to discontinuation of carfilzomib | 5 | 20

3. Secondary Outcome: Overall Survival
Description: Since participants were only followed up to 30 days after administration of last dose of study drug per protocol, Kaplan-Meier estimates of overall survival were not calculated. The number of participants who died within 30 days after administration of last dose of study drug is reported.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of carfilzomib after enrollment in PX-171-010.
Measure: Number; unit: participants
Arm/Group | Solid Tumors | Multiple Myeloma
Number analyzed (Participants) | 9 | 91
participants | 1 | 7

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time between the start of treatment and first evidence of documented disease progression or death (due to any cause), whichever occurred first.
  Disease progression was determined by the local investigator for regimens with the same baseline using the International Uniform Response Criteria (IMWG-URC) for participants with multiple myeloma and Response Evaluation Criteria in Solid Tumors (RECIST) criteria for solid tumor participants.
  PFS was re-calculated whenever the baseline was reset due to addition of new anti-cancer therapy or increase of carfilzomib dose/frequency.
Time Frame: From first dose of study drug in study PX-171-010 to 30 days after the last dose; median duration of treatment was 14 weeks for participants with solid tumors and 44 weeks for participants with multiple myeloma.
Population: Enrolled participants excluding those with no postbaseline endpoint data subsequent to at least 1 dose of the study drug on the PX-171-010 protocol and participants who lacked baseline data for those analyses that required baseline data. Only participants with regimens that continued from the initial study without baseline being reset are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Solid Tumors | Multiple Myeloma
Number analyzed (Participants) | 6 | 58
months | 41.9 [NA to NA] — In this cohort participants were not followed until confirmed progressive disease. Only one participant was followed until an event; therefore PFS data were not mature and confidence interval could not be calculated. | 19.6 [10.2 to 30.6]

5. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) was defined as the time between start of treatment to the first documentation of disease progression. TTP was re-calculated whenever the baseline was reset due to addition of new anti-cancer therapy or increase of carfilzomib dose/frequency.
Time Frame: as for outcome 4
Population: Enrolled participants excluding those with no postbaseline endpoint data subsequent to at least 1 dose of the study drug on the PX-171-010 protocol and participants who lacked baseline data for those analyses that required baseline data Only participants with regimens that continued from the initial study without baseline being reset are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Solid Tumors | Multiple Myeloma
Number analyzed (Participants) | 6 | 58
months | NA [NA to NA] — Could not be estimated due to the low number of events | 19.6 [10.2 to 30.6]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after the last dose; median duration of treatment was 14 weeks for participants with solid tumors and 44 weeks for participants with multiple myeloma.
Description: The protocol indicated that AEs leading to dose modification, dose discontinuation, CTCAE grade 3+, serious AEs and all-grade peripheral neuropathy AEs were collected in the study.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Solid Tumors | Multiple Myeloma
All-Cause Mortality (participants affected / at risk) | 1/9 | 7/91
Serious Adverse Events (participants affected / at risk) | 5/9 | 57/91
Other Adverse Events (participants affected / at risk) | 6/9 | 69/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Solid Tumors (N=9) | Multiple Myeloma (N=91)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 5
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 2
Infusion related reaction (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 3
Catheter sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Haemophilus sepsis (Infections and infestations) | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 6
Intraspinal abscess (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 10
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 2
Pneumonia viral (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Solid Tumors (N=9) | Multiple Myeloma (N=91)
Anaemia (Blood and lymphatic system disorders) | 0 | 18
Neutropenia (Blood and lymphatic system disorders) | 0 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 16
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 12
Nausea (Gastrointestinal disorders) | 2 | 11
Vomiting (Gastrointestinal disorders) | 3 | 5
Asthenia (General disorders) | 1 | 1
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 3 | 16
Infusion site pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 4
Sensation of pressure (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 0 | 6
Sinusitis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 21
Urinary tract infection (Infections and infestations) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 7
Dysarthria (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 10
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 3
Dysuria (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 14
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2011-03-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT00884312/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT00884312/SAP_001.pdf